CLINICAL TRIAL: NCT03279393
Title: Stress and Atherosclerotic Plaque Macrophages: A Systems Biology Approach - PET/MRI of the Brain-hematopoiesis-atherosclerosis Axis in PTSD Patients
Brief Title: PPG Project 3 - PET/MRI of the Brain-hematopoiesis-atherosclerosis Axis in PTSD Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zahi Fayad (Other)
Collaborators: Massachusetts General Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Zahi Fayad, Director of Translational and Molecular Imaging Institute, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GCO 15-0893 P3; 1P01HL131478 (NIH)
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: PTSD; Trauma; Healthy
Keywords: Post-Traumatic Stress Disorder; PTSD; trauma; stress; atherosclerosis; macrophage; plaque burden; vascular inflammation; atherosclerotic inflammation; PET/MRI; 18F-FDG-PET
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Atherosclerosis | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PTSD Subjects (Active Comparator)
  Interventions: Drug: fluorodeoxyglucose (FDG)-PET/MRI
- Trauma Control Subjects (Active Comparator)
  Interventions: Drug: fluorodeoxyglucose (FDG)-PET/MRI
- Healthy Control Subjects (Placebo Comparator)
  Interventions: Drug: fluorodeoxyglucose (FDG)-PET/MRI

INTERVENTIONS:
Drug: fluorodeoxyglucose (FDG)-PET/MRI — Innovative PET combined with magnetic resonance imaging (PET/MRI) to simultaneously study the hematopoietic system, the artery wall, and the brain's fear system, which comprises the amygdala and anterior cingulate cortex (ACC)

SUMMARY:
Project 3 of the PPG grant "Stress and Atherosclerotic Plaque Macrophages A Systems Biology Approach," funded by the NHLBI, examines the relationship between psychosocial stress and atherosclerotic inflammation, cell proliferation and burden using novel PET/MRI. Individuals with post-traumatic stress disorder, trauma controls and healthy controls will be recruited into a two-center clinical study. The study team will use functional MRI to examine the relationship between activation of fear circuits in the brain and relate these data to hematopoietic system activation, and vascular inflammation measured by FDG-PET, and atherosclerotic burden measured by MRI.

DETAILED DESCRIPTION:
In Project 3, the study team will employ innovative PET combined with magnetic resonance imaging (PET/MRI) to simultaneously study the hematopoietic system, the artery wall, and the brain's fear system, which comprises the amygdala and anterior cingulate cortex (ACC), to elucidate the relationship between psychosocial stress and systemic inflammation/atherosclerosis in a two center clinical study looking at: I) individuals with PTSD, II) individuals without PTSD but with exposure to severe psychosocial trauma (Trauma Control), and III) matched volunteers with neither PTSD nor exposure to trauma (Healthy Control). Participants in the three study groups, recruited from urban settings in New York and Boston, will be group-matched by age, gender, and Framingham risk scores (FRS). The study team will recruit 80 subjects in each group and in Aim 1, investigate the relationship between PTSD and atherosclerotic inflammation and burden measured by PET/MRI. In Aim 2, the study team will examine the relationships between brain's fear circuit responsiveness to threat assessed by functional MRI (fMRI) and white matter integrity assessed by diffusion tensor imaging (DTI) and relate these data to hematopoietic system activation, and vascular inflammation measured by fluorodeoxyglucose (FDG)-PET and atherosclerotic burden measured by MRI.

The following will occur during the imaging visit:

1. Questionnaire: study staff will administer a standardized questionnaire to collect general information on age, gender, race, and current contact information. A PET/MRI pre-screening form will also be administered to confirm eligibility for the PET/MRI scan. This questionnaire is specific to the PET/MRI scan.
2. Blood pressure: One blood pressure reading, taken in the dominant arm, will be performed per the American Heart Association recommendations.
3. Anthropometrics: Body weight and height will be measured according to standard methods and body mass index will be calculated as an index for obesity. Waist circumference will also be measured.
4. Blood draw: approximately 3 tablespoons of blood will be drawn to evaluate clinical variables.
5. Imaging at Mount Sinai or Massachusetts General Hospital: A Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI) scan
6. Urine drug screen
7. C-SSRS safety assessment

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Group 1 (PTSD Subjects)

* Male or female aged 30-65 years;
* Meets DSM-V criteria for Post-Traumatic Stress Disorder (PTSD) from at least one year prior to enrollment (as assessed using the SCID and the CAPS);
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.

Inclusion for Group 2 (Trauma Control Subjects)

* Male or female aged 30-65 years;
* Meets DSM-V criteria A of Post-Traumatic Stress Disorder (PTSD) from at least one year prior to enrollment, without satisfying criteria for a PTSD diagnoses according to the DSM-V (as assessed using the SCID);
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.

Inclusion criteria for Group 3 (Healthy Control Subjects)

* Male or female aged 30-65 years;
* Does not meet for any current or past psychiatric diagnoses as defined by DSM-V criteria;
* Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.

Exclusion Criteria:

* Clinical history of atherosclerotic disease (prior myocardial infarction, stroke, peripheral artery disease)
* Clinical history or presence of significant central nervous system and neurological diseases (e.g., TBI, multiple sclerosis)
* History of class 3 or 4 heart failure, severe life-threatening arrhythmia (e.g., ventricular tachycardia) or severe mitral or aortic valvular disease Current, primary psychiatric disorder other than PTSD (not including ADD, ADHD)
* History or current schizophrenia or primary psychotic disorders (e.g. schizophrenia, schizoaffective disorder)
* Suicidal ideation with any intent or plan as measured by a Columbia Suicide Severity Rating Scale [C-SSRS] score of greater than 3 during the past month at the time of screening
* Current or history of a major cognitive disorder or evidence of cognitive impairment as assessed by a score of the Mini Mental Status Exam (MMSE) of <24
* Substance Use Disorder within the past 6 months;
* Hypnotic medications used PRN are allowed except within 24 hours of the scan assessment day (V1)
* Benzodiazepine medications used PRN (not to exceed 2 mg of lorazepam daily) are allowed except within 12 hours of the scan assessment day (V1)
* Positive urine-toxicology (u-tox) screening for illicit substances at assessment day
* Alcohol consumption above the NIAA cut-off for moderate alcohol intake (maximum 14 drinks for men and 7 drinks for women per week)
* Concomitant use of high intensity statins (atorvastatin ≥ 40 mg/day; rosuvastatin > 20 mg/day; pitavastatin ≥ 2 mg/day)
* Concomitant systemically-administered anti-inflammatory agents for chronic inflammatory conditions (e.g., methotrexate or anti-inflammatory biologics). On the other hand, NSAIDS, aspirin, and topical or inhaled steroids are permitted;
* Chronic inflammatory conditions including but not limited to psoriasis and rheumatoid arthritis;
* Subjects with malignancies that are within 5 years of remission are excluded.
* Clinically significant abnormalities of laboratories or advanced systemic disease (i.e. malignancy); specific cutoffs include:
* A value of >52 for high-sensitivity troponin (however a value between 13 and 52 will need PI clearance); a threshold of .03 and .01 respectively, for older generation troponin

  * Leukopenia: WBC <4.0
  * HsCRP >10
  * EGFR <60
  * Known or active liver disease with AST/ALT >3 times the ULN, Bil >2 times the ULN
  * Coagulation abnormalities such as INR >1.1, aPTT >34.9 (unless subject is on anticoagulation therapy)
* Type 1 diabetes
* Type 2 diabetes AND HbA1C > 7.5;
* Women who are pregnant;
* Any contraindications to MRI, including claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, and inability to lie still for 1 hour or more.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Atherosclerotic burden in PTSD using PET/MRI | Day 1
  The atherosclerosis burden as measured by 18F-FDG-PET/MRI

SECONDARY OUTCOMES:
Degree of brain fear circuit activation | Day 1
  The degree of brain fear circuit activation (both at rest and in response to validated stimuli) to be associated with activation of hematopoietic organs 18F-FDG PET imaging.
Level of circulating HPSCs | Day 1
Level of circulating immune cells | Day 1
Level of soluble inflammation biomarkers | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Zahi Fayad, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
After each imaging visit, de-identified images of the subject will be transferred via a secure BrickFTP server to the Coordinating Center (Icahn School of Medicine at Mount Sinai) for storage and analysis.

REFERENCES:
- [Background] Fuster V, Kovacic JC. Acute coronary syndromes: pathology, diagnosis, genetics, prevention, and treatment. Circ Res. 2014 Jun 6;114(12):1847-51. doi: 10.1161/CIRCRESAHA.114.302806. Epub 2014 May 13. No abstract available. PMID 24824094
- [Background] Fuster V, Stein B, Ambrose JA, Badimon L, Badimon JJ, Chesebro JH. Atherosclerotic plaque rupture and thrombosis. Evolving concepts. Circulation. 1990 Sep;82(3 Suppl):II47-59. PMID 2203564
- [Background] Hansson GK, Libby P. The immune response in atherosclerosis: a double-edged sword. Nat Rev Immunol. 2006 Jul;6(7):508-19. doi: 10.1038/nri1882. Epub 2006 Jun 16. PMID 16778830
- [Background] Heidt T, Sager HB, Courties G, Dutta P, Iwamoto Y, Zaltsman A, von Zur Muhlen C, Bode C, Fricchione GL, Denninger J, Lin CP, Vinegoni C, Libby P, Swirski FK, Weissleder R, Nahrendorf M. Chronic variable stress activates hematopoietic stem cells. Nat Med. 2014 Jul;20(7):754-758. doi: 10.1038/nm.3589. Epub 2014 Jun 22. PMID 24952646
- [Background] Brudey C, Park J, Wiaderkiewicz J, Kobayashi I, Mellman TA, Marvar PJ. Autonomic and inflammatory consequences of posttraumatic stress disorder and the link to cardiovascular disease. Am J Physiol Regul Integr Comp Physiol. 2015 Aug 15;309(4):R315-21. doi: 10.1152/ajpregu.00343.2014. Epub 2015 Jun 10. PMID 26062635
- [Background] Plantinga L, Bremner JD, Miller AH, Jones DP, Veledar E, Goldberg J, Vaccarino V. Association between posttraumatic stress disorder and inflammation: a twin study. Brain Behav Immun. 2013 May;30:125-32. doi: 10.1016/j.bbi.2013.01.081. Epub 2013 Feb 4. PMID 23379997
- [Background] Nahrendorf M, Swirski FK. Lifestyle effects on hematopoiesis and atherosclerosis. Circ Res. 2015 Feb 27;116(5):884-94. doi: 10.1161/CIRCRESAHA.116.303550. PMID 25722442
- [Background] Edmondson D, Kronish IM, Shaffer JA, Falzon L, Burg MM. Posttraumatic stress disorder and risk for coronary heart disease: a meta-analytic review. Am Heart J. 2013 Nov;166(5):806-14. doi: 10.1016/j.ahj.2013.07.031. Epub 2013 Sep 24. PMID 24176435
- [Background] Thakur GS, Daigle BJ Jr, Dean KR, Zhang Y, Rodriguez-Fernandez M, Hammamieh R, Yang R, Jett M, Palma J, Petzold LR, Doyle FJ 3rd. Systems biology approach to understanding post-traumatic stress disorder. Mol Biosyst. 2015 Apr;11(4):980-93. doi: 10.1039/c4mb00404c. PMID 25627823
- [Background] Graebe M, Borgwardt L, Hojgaard L, Sillesen H, Kjaer A. When to image carotid plaque inflammation with FDG PET/CT. Nucl Med Commun. 2010 Sep;31(9):773-9. doi: 10.1097/MNM.0b013e32833c365e. PMID 20543757
- [Background] Tawakol A, Fayad ZA, Mogg R, Alon A, Klimas MT, Dansky H, Subramanian SS, Abdelbaky A, Rudd JH, Farkouh ME, Nunes IO, Beals CR, Shankar SS. Intensification of statin therapy results in a rapid reduction in atherosclerotic inflammation: results of a multicenter fluorodeoxyglucose-positron emission tomography/computed tomography feasibility study. J Am Coll Cardiol. 2013 Sep 3;62(10):909-17. doi: 10.1016/j.jacc.2013.04.066. Epub 2013 May 30. PMID 23727083
- [Background] Calcagno C, Cornily JC, Hyafil F, Rudd JH, Briley-Saebo KC, Mani V, Goldschlager G, Machac J, Fuster V, Fayad ZA. Detection of neovessels in atherosclerotic plaques of rabbits using dynamic contrast enhanced MRI and 18F-FDG PET. Arterioscler Thromb Vasc Biol. 2008 Jul;28(7):1311-7. doi: 10.1161/ATVBAHA.108.166173. Epub 2008 May 8. PMID 18467641
- [Background] Hodes GE, Pfau ML, Leboeuf M, Golden SA, Christoffel DJ, Bregman D, Rebusi N, Heshmati M, Aleyasin H, Warren BL, Lebonte B, Horn S, Lapidus KA, Stelzhammer V, Wong EH, Bahn S, Krishnan V, Bolanos-Guzman CA, Murrough JW, Merad M, Russo SJ. Individual differences in the peripheral immune system promote resilience versus susceptibility to social stress. Proc Natl Acad Sci U S A. 2014 Nov 11;111(45):16136-41. doi: 10.1073/pnas.1415191111. Epub 2014 Oct 20. PMID 25331895
- [Background] Kim EJ, Kim S, Kang DO, Seo HS. Metabolic activity of the spleen and bone marrow in patients with acute myocardial infarction evaluated by 18f-fluorodeoxyglucose positron emission tomograpic imaging. Circ Cardiovasc Imaging. 2014 May;7(3):454-60. doi: 10.1161/CIRCIMAGING.113.001093. Epub 2014 Jan 31. PMID 24488982
- [Background] Shin LM, Lasko NB, Macklin ML, Karpf RD, Milad MR, Orr SP, Goetz JM, Fischman AJ, Rauch SL, Pitman RK. Resting metabolic activity in the cingulate cortex and vulnerability to posttraumatic stress disorder. Arch Gen Psychiatry. 2009 Oct;66(10):1099-107. doi: 10.1001/archgenpsychiatry.2009.138. PMID 19805700